CLINICAL TRIAL: NCT00201981
Title: Rebamipide Ophthalmic Suspension in the Treatment of Dry Eye: A Multicenter, Phase 3, Randomized, Double-Masked, Placebo-Controlled, Parallel-Group, 52 Week Study
Brief Title: Study of Rebamipide Eye Drops to Treat Dry Eye
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Collaborators: Novartis (Industry)
Responsible Party: Juan Guzman, MD/ Sr. Director, Global Clinical Development, Otsuka Pharmaceutical Development & Commercialization
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 37E-03-202
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2008-01-07 (Estimated); Status verified 2008-01

CONDITIONS: Keratoconjunctivitis Sicca
Keywords: dry eye; keratoconjunctivitis sicca
MeSH Terms: conditions — Keratoconjunctivitis Sicca; Dry Eye Syndromes | interventions — rebamipide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (3):
- 1 (Active Comparator): rebamipide 1%
  Interventions: Drug: Rebamipide
- 2 (Active Comparator): Rebamipide 2%
  Interventions: Drug: Rebamipide
- 3 (No Intervention): placebo

INTERVENTIONS:
Drug: Rebamipide — 1. OPC as a single drop per eye (approx 50 µL) 4 times per day for 52 weeks
  2. OPC as a single drop per eye (approx 50 µL) 4 times per day for 52 weeks
  Arms: 1; 2

SUMMARY:
The purpose of this study is to determine the potential safety and effectiveness of rebamipide eye drops, an investigational eye drop being developed for the treatment of keratoconjunctivitis sicca (dry eye).

DETAILED DESCRIPTION:
There is a need for effective therapy for dry eye that treats the underlying cause of the syndrome. The goal of this study is to assess the impact of rebamipide on dry eye symptom.

ELIGIBILITY:
Inclusion Criteria:

* must have symptoms of dry eye for a minimum of 6 months
* must be able to sign and date an informed consent

Exclusion Criteria:

* presence of anterior segment disease
* glaucoma or ocular hypertension
* using Restasis
* use of topically instilled ocular medications during study
* use of contact lenses
* history of ocular surgery within 12 months
* females who are pregnant, breast feeding, or child-bearing potential and not willing to remain abstinent or use contraception
* presence of Stevens-Johnson syndrome
* any anticipated change in medication through-out study
* concurrent involvement in another study or previous receipt of this drug
* cannot be safely be weaned off of ocular medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 740 (Estimated)
Dates: Start 2004-05; Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
fluorescein corneal staining (FCS) total score at week 12 and the average primary ocular discomfort (POD) severity score at week 12 | 12 week and 26 week

SECONDARY OUTCOMES:
fluorescein corneal staining (FCS) total score at week 26 and the average primary ocular discomfort (POD) severity score at week 26 | 12 week and 26 week

CONTACTS AND LOCATIONS:
Overall Officials: Gary Foulks, MD, Study Chair — University of Louisville
Locations (63):
- United States (63):
  - Alabama Research Center, LLC, Birmingham, Alabama
  - Sun Valley Arthritis Center, Ltd., Glendale, Arizona
  - Pivotel Research Center, Peoria, Arizona
  - Hope research Institute, Phoenix, Arizona
  - Buena Vista Eye Care Center, Phoenix, Arizona
  - Radiant Research, Scottsdale, Arizona
  - Sall Eye Research Center, Artesia, California
  - Radiant Research - Irvine, Irvine, California
  - Scripps Clinic Medical Group, Inc., La Jolla, California
  - American Eye Institute, Los Angeles, California
  - Eye Clinic of San Diego, San Diego, California
  - Healthcare Partners Medical Group, Torrance, California
  - Centennial Eye Associates, Centennial, Colorado
  - Corneal Consultants of Colorado, Littleton, Colorado
  - Western States Clinical Research, Inc., Wheat Ridge, Colorado
  - Peter C. Donshik, MDPC, Bloomfield, Connecticut
  - Opticare Eye Health Center, Waterbury, Connecticut
  - The Eye Associates, Bradenton, Florida
  - Hernando Eye Institute, Brooksville, Florida
  - Radiant Research, Inc. - Lake Worth, Lake Worth, Florida
  - Suncoast Clinical Research, Inc., New Port Richey, Florida
  - Eye Associates International, Ormond Beach, Florida
  - Pinellas Eye Center, Pinellas Park, Florida
  - Ft. Lauderdale Eye Institute, Sunrise, Florida
  - Marvin E. Greenberg, MD PA 7, Tamarac, Florida
  - Clinical Research of West Florida, Inc., Tampa, Florida
  - International Eye Center, Tampa, Florida
  - Omni Eye Services, Atlanta, Georgia
  - University of Kentucky, Department of Ophthamology, Lexington, Kentucky
  - Kentucky Lions Eye Center, Louisville, Kentucky
  - Gulf Coast Research Associates, Inc., Baton Rouge, Louisiana
  - Danial Long, MD, Gretna, Louisiana
  - Lakeview Optical, New Orleans, Louisiana
  - Eye Center Northeast, Bangor, Maine
  - Krieger Eye Institute, Baltimore, Maryland
  - The Wilmer Eye Institute, Lutherville, Maryland
  - New England Eye Center, Boston, Massachusetts
  - The Eye Institute - Lahey Clinic North, Peabody, Massachusetts
  - Mississippi Eye Associates, Ocean Springs, Mississippi
  - Montana Medical Research, LLC, Missoula, Montana
  - Clinical Research Center of Nevada, Las Vegas, Nevada
  - Eye Associates of New Mexico, Albuquerque, New Mexico
  - Western New York Eye Center, Orchard Park, New York
  - Glaucoma Consultants of the Capital Region, Slingerlands, New York
  - Orellana Retina Associates, PLLC, Raleigh, North Carolina
  - University Hospitals of Cleveland, Cleveland, Ohio
  - Comprehensive Opthalmology & Optical Services, Cleveland, Ohio
  - Clinical Research Source, Inc., Perryberg, Ohio
  - Clinical Research Institute of Southern Oregon, Medford, Oregon
  - Northwest Corneal Services, Portland, Oregon
  - Vision Surgery and Laser Center, Roseburg, Oregon
  - West Hills Vision Center, Moon Township, Pennsylvania
  - Glaucoma Consultants and Center for Eye Research, Mt. Pleasant, South Carolina
  - University Eye Surgeons, Maryville, Tennessee
  - St. Luke's Eye Institute, Amarillo, Texas
  - Eye Clinic of Austin, Austin, Texas
  - Baylor College of Medicine, Houston, Texas
  - Surgical Eye Associates, PA, Houston, Texas
  - Brazosport Eye Institute, Lake Jackson, Texas
  - Axia Research, Salt Lake City, Utah
  - John Moran Eye Center, University of Utah, Salt Lake City, Utah
  - Physicians Research Options, LC, Sandy City, Utah
  - Access Eye Research Center, Fredericksburg, Virginia

REFERENCES:
- [Background] Yamasaki K, Ishiyama H, Imaizumi T, Kanbe T, Yabuuchi Y. Effect of OPC-12759, a novel antiulcer agent, on chronic and acute experimental gastric ulcer, and gastric secretion in rats. Jpn J Pharmacol. 1989 Apr;49(4):441-8. doi: 10.1254/jjp.49.441. PMID 2542684
- [Background] Yamasaki K, Kanbe T, Chijiwa T, Ishiyama H, Morita S. Gastric mucosal protection by OPC-12759, a novel antiulcer compound, in the rat. Eur J Pharmacol. 1987 Oct 6;142(1):23-9. doi: 10.1016/0014-2999(87)90649-2. PMID 3480223
- [Background] Yoshikawa T, Naito Y, Tanigawa T, Kondo M. Free radical scavenging activity of the novel anti-ulcer agent rebamipide studied by electron spin resonance. Arzneimittelforschung. 1993 Mar;43(3):363-6. PMID 8387788
- [Background] Yoshikawa T, Naito Y, Nakamura S, Nishimura S, Kaneko T, Iinuma S, Takahashi S, Kondo M, Yamasaki K. Effect of rebamipide on lipid peroxidation and gastric mucosal injury induced by indometacin in rats. Arzneimittelforschung. 1993 Dec;43(12):1327-30. PMID 8141822
- [Background] Yamasaki K, et al. Effect of OPC 12759 on the production of oxygen-derived free radical from human polymorphonuclear leukocytes. In-house Report No. 004272.
- [Background] Yamasaki K, et al. Effect of OPC 12759 on gastric mucosal blood flow in rats-determination by the hydrogen gas clearance method. In-house Report No. 003915.
- [Background] Imaizumi, T, et al. Effect of OPC 12759 and cetraxate on gastric mucosal hemodynamics and oxygen sufficiency in rats-analysis by reflectance spectrophotometry. In-house Report No. 004101.
- [Background] Garcher C, Bron A, Baudouin C, Bildstein L, Bara J. CA 19-9 ELISA test: a new method for studying mucus changes in tears. Br J Ophthalmol. 1998 Jan;82(1):88-90. doi: 10.1136/bjo.82.1.88. PMID 9536889
- [Background] Danjo Y, Watanabe H, Tisdale AS, George M, Tsumura T, Abelson MB, Gipson IK. Alteration of mucin in human conjunctival epithelia in dry eye. Invest Ophthalmol Vis Sci. 1998 Dec;39(13):2602-9. PMID 9856770
- [Background] Pflugfelder SC, Tseng SC, Yoshino K, Monroy D, Felix C, Reis BL. Correlation of goblet cell density and mucosal epithelial membrane mucin expression with rose bengal staining in patients with ocular irritation. Ophthalmology. 1997 Feb;104(2):223-35. doi: 10.1016/s0161-6420(97)30330-3. PMID 9052626
- [Background] Kinoshita S, Kiorpes TC, Friend J, Thoft RA. Goblet cell density in ocular surface disease. A better indicator than tear mucin. Arch Ophthalmol. 1983 Aug;101(8):1284-7. doi: 10.1001/archopht.1983.01040020286025. PMID 6882259
- [Background] Rivas L, Oroza MA, Perez-Esteban A, Murube-del-Castillo J. Morphological changes in ocular surface in dry eyes and other disorders by impression cytology. Graefes Arch Clin Exp Ophthalmol. 1992;230(4):329-34. doi: 10.1007/BF00165940. PMID 1505763
- [Background] Nelson JD, Wright JC. Conjunctival goblet cell densities in ocular surface disease. Arch Ophthalmol. 1984 Jul;102(7):1049-51. doi: 10.1001/archopht.1984.01040030851031. PMID 6378156
- [Background] Ferris FL 3rd, Kassoff A, Bresnick GH, Bailey I. New visual acuity charts for clinical research. Am J Ophthalmol. 1982 Jul;94(1):91-6. PMID 7091289
- [Background] Lemp MA. Report of the National Eye Institute/Industry workshop on Clinical Trials in Dry Eyes. CLAO J. 1995 Oct;21(4):221-32. No abstract available. PMID 8565190
- [Background] Gail M, Simon R. Testing for qualitative interactions between treatment effects and patient subsets. Biometrics. 1985 Jun;41(2):361-72. PMID 4027319
- [Background] Davis CS, Chung Y. Randomization model methods for evaluating treatment efficacy in multicenter clinical trials. Biometrics. 1995 Sep;51(3):1163-74. PMID 7548700